CLINICAL TRIAL: NCT01392976
Title: A Phase I, Open-Label, Two-stage, Randomized, Crossover, Comparative Pharmacokinetic and Safety Study of Two Formulations of CO-1.01 for Injection in Patients With Advanced Solid Tumors
Brief Title: Safety and Pharmacokinetic Profiles of Two Formulations of CO-1.01 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CO-101-004
Record Dates: First submitted 2011-04-13; First posted 2011-07-13 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Advanced Solid Tumor
Keywords: cancer; advanced; solid; tumor; gemcitabine; human equilibrative nucleoside transporter-1 (hENT1); CO-1.01; CO-101; CO101
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CO-1.01 Formulation B (Experimental)
  Interventions: Drug: CO-1.01 Formulation B (Aqueous suspension containing 30 mg/mL of drug solubilized in purified phospholipids)
- CO-1.01 Formulation A (Active Comparator)
  Interventions: Drug: CO-1.01 Formulation A (Aqueous suspension containing 15 mg/mL of drug solubilized in purified phospholipids)

INTERVENTIONS:
Drug: CO-1.01 Formulation A (Aqueous suspension containing 15 mg/mL of drug solubilized in purified phospholipids) — 1250 mg/m2 intravenous infusion on Day 1 for Treatment Sequence 1 and Day 8 for Treatment Sequence 2.
  Arms: CO-1.01 Formulation A
Drug: CO-1.01 Formulation B (Aqueous suspension containing 30 mg/mL of drug solubilized in purified phospholipids) — 1250 mg/m2 intravenous infusion on Day 1 for Treatment Sequence 2 and Day 8 for Treatment Sequence 1.
  Arms: CO-1.01 Formulation B

SUMMARY:
The purpose of this study is to compare the pharmacokinetic and safety profiles of two formulations of CO-1.01 in patients with Advanced Solid Tumors.

DETAILED DESCRIPTION:
Gemcitabine is used alone or in combination with other chemotherapy as a treatment for several solid tumor types, including pancreatic cancer, NSCLC, and ovarian cancer. Unfortunately, many patients fail to derive benefit from this treatment. No clinical or molecular marker has been established to predict benefit from gemcitabine therapy, so patients are treated empirically until evidence of disease progression or worsening performance status.

The potential for human equilibrative nucleoside transporter-1 (hENT1) expression to predict survival in gemcitabine-treated patients has been studied, and data suggest that patients with low levels of tumor cell hENT1 expression derive less benefit from gemcitabine treatment than patients with high levels of tumor cell hENT1 expression. Furthermore, the PK profiles of CO-1.01 and gemcitabine are different, and this may also favorably influence the in vivo antiproliferative effects of CO-1.01. These data support the hypothesis that patients expressing low levels of hENT1 will derive minimal benefit from gemcitabine, but will receive benefit from CO-1.01 (gemcitabine elaidate) which enters tumor cells in a hENT1-independent fashion.

The formulation of CO-1.01 that is currently used in clinical studies contains 15 mg/mL of gemcitabine-5'-elaidate solubilized in purified phospholipids. Recently, Clovis Oncology developed a 30 mg/ml formulation which will be characterized in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with a histologically confirmed solid tumor malignancy that is metastatic or unresectable for which there is no standard curative or palliative treatment option available and for which CO-1.01 treatment would be appropriate
* Life expectancy of at least 3 months
* Performance status (ECOG)0 or 1
* Age ≥18 years
* Adequate hematological and biological function
* Written consent on an Institutional Review Board/Independent Ethics Committee-approved IC Form prior to any study-specific evaluation

Exclusion Criteria:

* Clinically significant abnormal 12-lead ECG or QTcF>450msec (males) or >470 msec (females), PR>240 msec, or a QRS>110msec
* Family history of long QT syndrome
* Implantable pacemaker or implantable cardioverter defibrillator
* Symptomatic brain metastases
* Concomitant treatment with prohibited medications
* Treatment with a previous regimen of CO-1.01 within 30 days or randomization
* Treatment with any medication known to produce QT prolongation
* Surgical procedures are not allowed ≥14 days prior to administration of CO-1.01. In all cases, the patient must be sufficiently recovered and stable
* History of allergy to gemcitabine or eggs
* Females who are pregnant or breastfeeding
* Refusal to use adequate contraception for fertile patients (females and males) for 6 months after the last dose of CO-1.01
* Presence of any serious of unstable concomitant systemic disorder incompatible with the clinical study (e.g., substance abuse, psychiatric disturbance, uncontrolled intercurrent illness including active infection, arterial thrombosis, and symptomatic pulmonary embolism)
* Any other reason the investigator considers the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Ratio of the AUC0-∞ of the two formulations of CO-1.01 given as a 30 min i.v. infusion at 1250 mg/m2 | Serum & urine PK sampling at multiple timepoints through Cycle 1: Day 1 & Day 8

SECONDARY OUTCOMES:
PK of CO-1.01 and metabolites in plasma and urine after 1250 mg/m2 CO-1.01 given as a single 30 min i.v. infusion | Serum & urine PK sampling at multiple timepoints through Cycle 1: Day 1 & Day 8
QT/QTc interval of the ECG | Continuous ECG monitoring 8 hrs pre & post dose C1: D1, D8. 12 lead ECGs pre-dose, 30mins, 24hr, 48hr, 72hr C1: D1, D8
Relationship between plasma concentration of CO-1.01 and QT/QTc interval of the ECG | Plasma: multiple timepoints through C1D1 and D8. ECG: continuous monitoring 8 hrs pre & post dose C1: D1, D8. 12 lead ECGs pre-dose, 30mins, 24hr, 48hr, 72hr C1:D1, D8.
Drug tolerability and toxicity using clinical AE monitoring and clinical laboratory testing | From the time of signing the ICF until 28 days after last dose of CO-101. CO-101 dosed on C1D1, C1D8, C1D15, C2D1, C2D8, and C2D15.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Schellens, MD PhD, Principal Investigator — The Netherlands Cancer Institute, Amsterdam, Netherlands
Locations (3):
- Netherlands (3):
  - The Netherlands Cancer Institute, Amsterdam
  - Maastricht University Medical Center, Maastricht
  - University Medical Center Utrecht, Utrecht